CLINICAL TRIAL: NCT00876499
Title: Relationship Among Fatigue, Symptoms, Melatonin and Sleep in PBT Patients Undergoing Radiation Therapy
Brief Title: Fatigue, Sleep and Cytokines in Primary Brain Tumor (PBT) Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0747
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Brain Cancer
Keywords: Primary Brain Tumor; PBT; Brain Cancer; Primary glioma; Astrocytoma; Oligodendroglioma; Oligo-astrocytoma; Ependymoma; Anaplastic astrocytoma; Anaplastic oligodendroglioma; Anaplastic oligo-astrocytoma; Anaplastic ependymoma; Fatigue; Cytokines; Questionnaires; Actigraphy; Sleep Disturbance; Radiation Therapy
MeSH Terms: conditions — Brain Neoplasms; Astrocytoma; Oligodendroglioma; Ependymoma; Fatigue; Parasomnias | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Questionnaire
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — A total of 8 questionnaires regarding fatigue taking approximately 30 minutes each, given before radiation therapy, weekly during, and after completion.
  Other Names: Survey

SUMMARY:
This goal of this research study is to learn more about fatigue, sleep quality, and other symptoms in patients with primary brain tumors who are being treated with radiation therapy.

Objectives:

PRIMARY OBJECTIVE:

1. The primary objective of this study is to provide preliminary data describing the severity and change over time in fatigue using the Brief Fatigue Inventory (BFI) during radiation therapy for patients with primary gliomas.

SECONDARY OBJECTIVES:

1. To evaluate longitudinal changes in the severity of symptoms and the mean symptom burden as measured by the M.D. Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT) and mood using the Profile of Mood States (POMS) during radiation therapy.
2. To assess alterations in circadian rhythms using actigraphy during radiation therapy and the association with sleep quality tools - Pittsburgh Sleep Quality Index (PSQI) and the Epworth Sleepiness Scale(ESS), and the severity of BFI and MDASI-BT scores over time.
3. To explore the association between the levels of salivary hormones (melatonin and cortisol) and the occurrence of fatigue and symptom burden.

DETAILED DESCRIPTION:
Questionnaires:

If you decide to take part in this study, before starting radiation therapy, weekly during radiation therapy, and again 3-4 weeks and 6-8 weeks after completing radiation therapy, you will complete 4 questionnaires. Three (3) of the questionnaires will be completed during a study visit, and the last 1 will be completed at home the next time you come into the clinic. You will return the questionnaire completed at home to the study doctor at a study visit. The questionnaires will ask questions about fatigue, any symptoms you may have, and your sleeping habits. It should take about 30 minutes total to complete all of the questionnaires each time.

Sleep Diary:

You will complete a sleep diary. The sleep diary will be provided to you before starting radiation therapy. You will record information in it about your sleep habits, caffeinated beverages and drugs you may take, the quality of your sleep, and how you feel when you wake up. You will complete the sleep diary during the 48 hours that you are wearing the actigraphy watch. You will bring the sleep diary to the clinic every week for the study doctor to review.

Actigraphy Watch:

You will wear an actigraphy watch on your wrist for 48 hours before starting radiation therapy, for 48 hours each week during radiation therapy, and again for 48 hours 3-4 weeks and 6-8 weeks after completing radiation therapy. The actigraphy watch will measure your activity during the day and night. You will bring the actigraphy watch to the clinic every week for the study doctor to review.

Saliva Collection:

You will collect a saliva sample four times during the day before starting radiation therapy, one time during the third and last week of radiation therapy, and again 3-4 weeks and 6-8 weeks after completing radiation therapy. These samples will be used to measure levels of neurotransmitters and hormone levels. These are substances which are released in the body that may affect sleep and the immune system.

Length of Study:

You will remain on study for about 8 weeks after you complete radiation therapy.

This is an investigational study. Up to 20 patients will take part in this study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. A new diagnosis of a primary glioma, astrocytoma, oligodendroglioma, oligo-astrocytoma, ependymoma, tanycytic ependymoma, anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic oligo-astrocytoma, anaplastic ependymoma
2. Radiation therapy as part of the plan of care
3. Age >/= 18 years of age. Children are excluded from this study because of differences in tumor location and biology with differing symptom clusters. A separate study will be conducted in the future with children.
4. Ability to speak, write, and read English
5. On corticosteroids at the initiation of radiation therapy.

Exclusion Criteria:

1. Tumors involving the suprasellar region, including the pituitary and hypothalamus
2. Cognitive deficits which limit ability to self-report symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals over 18 years of age with a primary brain tumor scheduled for radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Patient Responses to Brief Fatigue Inventory (BFI) | BFI at baseline, at each weekly assessment, and again at the post-therapy assessment (3-4 weeks following chemotherapy).

CONTACTS AND LOCATIONS:
Overall Officials: Mark R. Gilbert, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org